CLINICAL TRIAL: NCT02633449
Title: Augmentation of Cognitive-Behavioral Psychotherapy With Prefrontal Direct Current Stimulation in Major Depression (Psychotherapy Plus)
Brief Title: Psychotherapy Plus: Combining Cognitive Behavioral Therapy With tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of München (Other); University Hospital Tuebingen (Other); University of Freiburg (Other); University of Leipzig (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Malek Bajbouj, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01EE1403F
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Major Depression
Keywords: tDCS; cognitive behavioral therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cognitive behavioral therapy + tDCS (Experimental): Group cognitive behavioral therapy combined with tDCS
  Interventions: Behavioral: cognitive behavioral therapy; Device: tDCS
- cognitive behavioral therapy + sham-tDCS (Active Comparator): Group cognitive behavioral therapy combined with sham-tDCS
  Interventions: Behavioral: cognitive behavioral therapy; Device: sham-tDCS
- cognitive behavioral therapy (Placebo Comparator): Group cognitive behavioral therapy only
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 12 sessions of group cognitive behavioral therapy, six patients, two therapists, duration: 100 minutes, two sessions per week for a total of six weeks
Device: tDCS — transcranial direct current stimulation during cognitive behavioral therapy with delayed onset after 10 minutes for 30 minutes, 1-2 mA, anode over electrode position F3, cathode over F4
  Arms: cognitive behavioral therapy + tDCS
Device: sham-tDCS — sham transcranial direct current stimulation during cognitive behavioral therapy with delayed onset after 10 minutes for 30 minutes, anode over electrode position F3, cathode over F4
  Arms: cognitive behavioral therapy + sham-tDCS

SUMMARY:
The study will investigate whether cognitive behavioral psychotherapy (CBT) combined with prefrontal transcranial direct current stimulation (tDCS) is more efficacious with regard to symptom reduction in depressed patients than CBT combined with sham-tDCS or CBT alone.

DETAILED DESCRIPTION:
Brain stimulation techniques are widely seen as promising treatment alternatives for patients not responding to or tolerating psychotropic medication. In particular, transcranial direct current stimulation (tDCS) is of special interest due to its potential to be used by a large number of patients because of its comparably ease of usage and good tolerability. Thus, a large number of studies investigating clinical effects of tDCS have been performed with statistically significant effects but that are of moderate clinical relevance. Clinical studies have mainly focused on the prefrontal cortex (PFC) as the main stimulation target based on findings of numerous studies indicating the lateral PFC to be a key dysfunctional node within brain networks involved in the pathophysiology of depression.

Studies in clinical and healthy participants indicate that tDCS is capable of positively augmenting prefrontal functions that are relevant for a successful cognitive behavioral therapy. More specifically, it has been shown that tDCS is capable of improving reappraisal strategies as well as the use of cognitive control techniques .

To date, previous studies have mainly addressed global antidepressant effects of tDCS and not effects on more circumscribed phenotypes mediated by top-down PFC processes such as impaired or biased emotional learning processes. All these trials have applied the stimulation to patients while being in a resting position. Nonetheless, recent neuropsychological studies indicate that tDCS effects appear to be "activity dependent", meaning that the stimulation effects are greater when the brain region being stimulated is simultaneously engaged in a cognitive task. Therefore, in the present study we will apply tDCS to patients with unipolar major depressive disorder during cognitive behavioral therapy (CBT), a well-established and highly effective psychotherapeutic treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

- unipolar major depressive disorder

Exclusion Criteria:

* neurological diseases or relevant psychiatric diseases other than major depressive disorder
* current medication other than SSRI or Mirtazapine
* manic episodes (lifetime)
* psychotic symptoms (lifetime)
* treatment with psychotherapy within the past 2 years
* treatment with electroconvulsive therapy (lifetime)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2016-02; Primary Completion 2019-11-15 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in depression severity as measured by Montgomery Asberg Depression Rating Scale (MADRS) | 6, 18 and 30 weeks after randomization
  MADRS ratings by trained clinicans, comparison between MADRS at baseline to MADRS post intervention, group comparison: treatment group vs. the two control interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité University Medicine Berlin, Department of Psychiatry and Psychotherapy, Berlin, Germany

REFERENCES:
- [Derived] Aust S, Brakemeier EL, Spies J, Herrera-Melendez AL, Kaiser T, Fallgatter A, Plewnia C, Mayer SV, Dechantsreiter E, Burkhardt G, Strauss M, Mauche N, Normann C, Frase L, Deuschle M, Bohringer A, Padberg F, Bajbouj M. Efficacy of Augmentation of Cognitive Behavioral Therapy With Transcranial Direct Current Stimulation for Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jun 1;79(6):528-537. doi: 10.1001/jamapsychiatry.2022.0696. PMID 35442431
- [Derived] Bajbouj M, Aust S, Spies J, Herrera-Melendez AL, Mayer SV, Peters M, Plewnia C, Fallgatter AJ, Frase L, Normann C, Behler N, Wulf L, Brakemeier EL, Padberg F. PsychotherapyPlus: augmentation of cognitive behavioral therapy (CBT) with prefrontal transcranial direct current stimulation (tDCS) in major depressive disorder-study design and methodology of a multicenter double-blind randomized placebo-controlled trial. Eur Arch Psychiatry Clin Neurosci. 2018 Dec;268(8):797-808. doi: 10.1007/s00406-017-0859-x. Epub 2017 Dec 6. PMID 29214483